CLINICAL TRIAL: NCT04769531
Title: Effects of Hip Joint Mobilizations and Strength Training on Pain, Physical Function and Dynamic Balance in Patients With Knee Osteoarthritis: A Randomized Control Trial
Brief Title: Hip Joint Mobilizations and Strength Training in Patients With Knee OA Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Osteo-arthritis; Musculoskeletal; lower extremity manual therapy; clinical trial Manual therapy; Resistance training; posture
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: It is a randomized control trial. Total 66 patients will be carry out, 22 in each of the three groups that include 2 patients as a drop out per group.
  There will be two interventional groups and one control group. Treatment will be allocated normally using random number sheet generated by statistician.
Who Masked: Participant
Masking Description: After enrolling the patient, informed consent will be taken from each taken. All patients will be blinded to the type of information to avoid biasness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hip Joint Mobilizations (Experimental): Hip joint mobilizations Hip strength training Knee exercises
  Interventions: Other: Hip Joint Mobilizations; Other: Hip joint Muscle strength training; Other: knee strengthening and flexibility exercises
- Hip & Knee Muscles strength training (Experimental): Hip strength training Knee exercises
  Interventions: Other: Hip joint Muscle strength training; Other: knee strengthening and flexibility exercises
- Knee Muscles strength training (Active Comparator): Knee exercises
  Interventions: Other: knee strengthening and flexibility exercises

INTERVENTIONS:
Other: Hip Joint Mobilizations — i. Anterior-posterior glide ii. Posterior-anterior glide iii. Caudal glide iv. Posterior-anterior glide with Abduction, flexion, and lateral rotation
  Arms: Hip Joint Mobilizations
Other: Hip joint Muscle strength training — i. Hip abduction in side-lying ii. Hip extension in the prone position iii. Sideways walk iv. Hip abduction in stand up position v. Hip hitching
  Arms: Hip & Knee Muscles strength training; Hip Joint Mobilizations
Other: knee strengthening and flexibility exercises — i. STRENGTHENING EXERCISES: Knee extension static quads set, terminal knee extension while standing up, sitting leg press, partial squat, step-ups.
  ii. STRETCHING EXERCISES:: stretching of the calf, hamstring, and quadriceps-femoris.
  iii. RANGE OF MOTION EXERCISES: Knee in mid-flexion to full-extension, Knee in mid-flexion to full-flexion:

SUMMARY:
Knee osteoarthritis has been ranked 11th highest contributor to non-fatal burdens in the world. Many research studies have discussed the relationship of hip muscle with knee joint stating that impaired hip strength can be a reason for knee pain. Furthermore, mobilization has been shown to be helpful in reducing pain, increasing range of motion and physical function in Osteoarthritis. Despite the evidence, there are very few studies that actually conducted clinical trials to test the effectiveness of mobilizations and strengthening of hip muscles in knee Osteoarthritis. Therefore our aim is to evaluate the effectiveness of hip joint mobilizations and strength training in knee osteoarthritis.

OBJECTIVE: To determine the effects of hip joint mobilizations and strengthening exercises, on pain, physical function and dynamic balance in patients with knee osteoarthritis (OA) using Visual analog scale, Knee injury and Osteoarthritis Outcome Score and four square step test.

METHODOLOGY: A randomized control trial will be conducted on 66 subjects with knee osteoarthritis and age 50 years will be enrolled in this study after screening by referring consultants. This study will be carried out at Physiotherapy OPD of DUHS, Civil hospital Karachi and Rabia Moon Memorial Institute of Neurosciences Trust. Subjects will be assessed at baseline and after 18 sessions using Visual analog scale, Knee injury and Osteoarthritis Outcome Score and square step test for pain, physical functioning and dynamic balance respectively. The subjects will be allocated into three groups through simple random sampling. Group A (joint mobilization group) will receive hip mobilization techniques, hip strengthening exercises along with the best available knee exercises while group B (hip muscles strengthening group) will receive hip-strengthening exercises with the best available knee exercises. Group C (knee strengthening group) will be receiving the best available knee treatment including exercises only. Patients will receive a total of 18 sessions, 5 treatment sessions per week for four successive weeks. The data will be entered and analyzed using SPPS version 21. Repeated mean one way ANOVA will be applied to measure VAS and KOOS scores within the group, for pairwise comparison between groups, Tukey's test will be applied. Chi-square will be applied for FSST scoring. A P-Value less than 0.5 will be considered significant.

DETAILED DESCRIPTION:
STUDY DESIGN:

A randomized control trial

STUDY SETTING:

The study will be carried out at an outpatient department of the Institute of Physical Medicine and Rehabilitation, Civil hospital and Rabia Moon Memorial Institute of Neurosciences Trust, Karachi

STUDY DURATION:

The duration of the study is 6 months after the approval of the synopsis. Each subject will receive a total of 18 sessions, 5 treatment sessions per week over the period of 4 weeks. Each treatment session accounts for 30-45 minutes.

STUDY POPULATION:

Subjects with knee osteoarthritis who fulfilled the following study inclusion and exclusion criteria:

INCLUSION CRITERIA

* Patients with unilateral or bilateral knee OA.
* Subjects of 50 years or above
* palpable bony enlargement
* Crepitus on knee motion
* morning stiffness for less than 30 minutes
* Kellgren and Lawrence scale: Grade 1-3

EXCLUSION CRITERIA

* Patients with spinal surgery
* lower extremity arthroplasty
* Severe joint contractures and bony deformities of the lower extremity
* Amputation of lower extremity
* Recent trauma to lower extremity
* A cortisone injection to the hip/ knee within the previous 30 days
* Patient having mechanical back pain .i.e. lumbosacral radiculopathy and sciatica
* Patient with lower extremity bony deformities either acquired or congenital
* Patient with advanced hip OA.
* Systemic arthritis or rheumatoid arthritis

SAMPLE SIZE:

Total 66 patients will be carried out, 22 in each group that include 2 patients as a drop out per group. Using PASS version 11 software, two independent sample t-test and 95% confidence interval 80% power of the test, mean ± S.D of VAS in group A is 4.67 ± 1.59 and group B is 3.6 ± 1.06. The calculated sample size is 27 per group. But due to the unavailability of patients, we will take 22 patients per group within 6 months.

SAMPLING TECHNIQUE:

Non- probability purposive sampling technique. Treatment will be allocated normally using a random number sheet generated by a statistician.

DATA COLLECTION PROCEDURE:

Data collection will begin right after the approval. Subjects fulfilling the inclusion criteria will be selected. Informed consent would be obtained after explaining the study objectives and procedure. Each enrolled patient will be randomly allocated using a computer-generated random number list in group A or group B or group C. All patients will be blinded to the type of intervention. The outcome measures would be used to collect data from all participants. The Visual analog scale for pain intensity, Knee injury and osteoarthritis outcome score for physical functions along with four-step square test for dynamic balance would be used and recorded. Outcome results would be obtained at the baseline before starting the treatment after 3 weeks as a follow-up and after 6 weeks after the completion of the study. The study will be carried out for 6 weeks. 18 sessions of 30-45 minutes will be given. Every attempt within ethical constraints will be made to obtain and record outcome data. If symptoms precipitate, subjects will be advised to use a hot pack or cold pack and prescribe an analgesic to control pain and discomfort.

STUDY VARIABLES

i DEPENDENT:

VAS, KOOS, FFST

ii. INDEPENDENT:

Age, gender, strengthening, mobilization

STATISTICAL ANALYSES:

For pair-wise comparison between groups, repeated mean one-way ANOVA will be applied and if there is any difference we will apply Tukey's test. For within-group, chi-square and repeated one-way ANOVA will be applied for FSST and VAS, KOOS respectively.

Baseline, midline and final readings will be taken for each group

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral knee OA.
* Subjects of 50 years or above
* palpable bony enlargement
* Crepitus on knee motion
* morning stiffness for less than 30 minutes
* Kellgren and Lawrence scale: Grade 1-3

Exclusion Criteria:

* Patients with spinal surgery
* lower extremity arthroplasty
* Severe joint contractures and bony deformities of lower extremity
* Amputation of lower extremity
* Recent trauma to lower extremity
* A cortisone injection to the hip/ knee within previous 30 days
* Patient having mechanical back pain .i.e. lumbosacral radiculopathy and sciatica
* Patient with lower extremity bony deformities either acquired or congenital
* Patient with advanced hip OA.
* Systemic arthritis or rheumatoid arthritis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | up to 6 weeks
  Visual analog scale (VAS) is a tool evaluating subjective attitudes that cannot be directly measurable, it has a good Test-retest reliability. This scoring range from 0 to 10 cm, Where 0 stands for no pain and 10 indicates worse possible pain.
Four step square test | up to 6 weeks
  Four square step tests is a tool for assessing the dynamic balance and mobility while standing. It also assess the fall risk.
Koos | up to 6 weeks
  The Knee Injury and Osteoarthritis Outcome Score is a PROM having five sub scales used for knee osteoarthritis (OA), it monitors the course of disease and final outcomes following interventions. Each subscale is scored from 0 (extreme problems) to 100 (no problems). It has high test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Mehwish, MSAPT, Principal Investigator — Dow University of Health Sciences; Shahzad Ali Syed, MSPT, Study Director — Dow University of Health Sciences; Aftab Ahmed Mirza Baig, MSAPT, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Mora JC, Przkora R, Cruz-Almeida Y. Knee osteoarthritis: pathophysiology and current treatment modalities. J Pain Res. 2018 Oct 5;11:2189-2196. doi: 10.2147/JPR.S154002. eCollection 2018. PMID 30323653
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Wallace IJ, Worthington S, Felson DT, Jurmain RD, Wren KT, Maijanen H, Woods RJ, Lieberman DE. Knee osteoarthritis has doubled in prevalence since the mid-20th century. Proc Natl Acad Sci U S A. 2017 Aug 29;114(35):9332-9336. doi: 10.1073/pnas.1703856114. Epub 2017 Aug 14. PMID 28808025
- [Background] Iqbal MN, Haidri FR, Motiani B, Mannan A. Frequency of factors associated with knee osteoarthritis. J Pak Med Assoc. 2011 Aug;61(8):786-9. PMID 22356003
- [Background] Ro DH, Lee J, Lee J, Park JY, Han HS, Lee MC. Effects of Knee Osteoarthritis on Hip and Ankle Gait Mechanics. Adv Orthop. 2019 Mar 24;2019:9757369. doi: 10.1155/2019/9757369. eCollection 2019. PMID 31019809
- [Background] A. Tanvi, R. Amrita, R. Deepak, P. Kopa. Comparison of effect of hip joint mobilization and hip joint muscle strengthening exercises with knee osteoarthritis. Scientific Research Journal of India. 2014;3
- [Background] Currier LL, Froehlich PJ, Carow SD, McAndrew RK, Cliborne AV, Boyles RE, Mansfield LT, Wainner RS. Development of a clinical prediction rule to identify patients with knee pain and clinical evidence of knee osteoarthritis who demonstrate a favorable short-term response to hip mobilization. Phys Ther. 2007 Sep;87(9):1106-19. doi: 10.2522/ptj.20060066. Epub 2007 Jul 3. PMID 17609333
- [Background] Cliborne AV, Wainner RS, Rhon DI, Judd CD, Fee TT, Matekel RL, Whitman JM. Clinical hip tests and a functional squat test in patients with knee osteoarthritis: reliability, prevalence of positive test findings, and short-term response to hip mobilization. J Orthop Sports Phys Ther. 2004 Nov;34(11):676-85. doi: 10.2519/jospt.2004.34.11.676. PMID 15609488
- [Background] Ahmad A, Daud M. A COMPARATIVE STUDY BETWEEN JOINT MOBILIZATION AND CONVENTIONAL PHYSIOTHERAPY IN KNEE OSTEOARTHRITIS. Int J Physio [Internet]. 2016Apr.8 [cited 2021Feb.2];3(2):159-62. Available from: https://www.ijphy.org/index.php/journal/article/view/207
- [Background] A. Tanvi, R. Amrita, R. Deepak, P. Kopa.Comparison of effect of hip joint mobilization and hip joint muscle strengthening exercises with knee osteoarthritis. Scientific Research J of Ind 2014;3(1)
- [Background] Santos TR, Oliveira BA, Ocarino JM, Holt KG, Fonseca ST. Effectiveness of hip muscle strengthening in patellofemoral pain syndrome patients: a systematic review. Braz J Phys Ther. 2015 May-Jun;19(3):167-76. doi: 10.1590/bjpt-rbf.2014.0089. Epub 2015 May 29. PMID 26039034
- [Background] Bennell KL, Hunt MA, Wrigley TV, Hunter DJ, McManus FJ, Hodges PW, Li L, Hinman RS. Hip strengthening reduces symptoms but not knee load in people with medial knee osteoarthritis and varus malalignment: a randomised controlled trial. Osteoarthritis Cartilage. 2010 May;18(5):621-8. doi: 10.1016/j.joca.2010.01.010. Epub 2010 Feb 6. PMID 20175973
- [Background] Schache MB, McClelland JA, Webster KE. Does the addition of hip strengthening exercises improve outcomes following total knee arthroplasty? A study protocol for a randomized trial. BMC Musculoskelet Disord. 2016 Jun 13;17:259. doi: 10.1186/s12891-016-1104-x. PMID 27295978
- [Background] Moore M, Barker K. The validity and reliability of the four square step test in different adult populations: a systematic review. Syst Rev. 2017 Sep 11;6(1):187. doi: 10.1186/s13643-017-0577-5. PMID 28893312
- [Background] Collins NJ, Prinsen CA, Christensen R, Bartels EM, Terwee CB, Roos EM. Knee Injury and Osteoarthritis Outcome Score (KOOS): systematic review and meta-analysis of measurement properties. Osteoarthritis Cartilage. 2016 Aug;24(8):1317-29. doi: 10.1016/j.joca.2016.03.010. Epub 2016 Mar 21. PMID 27012756
- [Background] Alviar MJ, Olver J, Brand C, Hale T, Khan F. Do patient-reported outcome measures used in assessing outcomes in rehabilitation after hip and knee arthroplasty capture issues relevant to patients? Results of a systematic review and ICF linking process. J Rehabil Med. 2011 Apr;43(5):374-81. doi: 10.2340/16501977-0801. PMID 21448553
- [Background] Gould D, Kelly D, Goldstone L, Gammon J. Examining the validity of pressure ulcer risk assessment scales: developing and using illustrated patient simulations to collect the data. J Clin Nurs. 2001 Sep;10(5):697-706. doi: 10.1046/j.1365-2702.2001.00525.x. PMID 11822520
- [Background] Hanrahan S, Van Lunen BL, Tamburello M, Walker ML. The Short-Term Effects of Joint Mobilizations on Acute Mechanical Low Back Dysfunction in Collegiate Athletes. J Athl Train. 2005 Jun;40(2):88-93. PMID 15970954
- [Background] Philadelphia Panel. Philadelphia Panel evidence-based clinical practice guidelines on selected rehabilitation interventions for knee pain. Phys Ther. 2001 Oct;81(10):1675-700. PMID 11589643
- [Background] Hengeveld E, Banks K.(ed) Maitland's Peripheral Manipulation. 4th ed. Elsevier: London.(2005)
- [Derived] Mehwish B, Ali SS, Mirza Baig AA. Effect of hip joint mobilisations and strength training on pain, physical function and dynamic balance in patients with Knee Osteoarthritis: A randomized controlled trial. J Pak Med Assoc. 2023 Apr;73(4):749-754. doi: 10.47391/JPMA.6223. PMID 37051976